CLINICAL TRIAL: NCT05574179
Title: Comparison of Sedative Effect of Dexmedetomidine and Midazolam for TIVA in Pediatric Population Undergoing Inguinal Hernia Repair, Randomized Controlled Trial
Brief Title: Comparison of Sedative Effect of Dexmedetomidine and Midazolam for TIVA
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheikh Zayed Medical College (Other Government)
Responsible Party: Principal Investigator, Barzah Durrani, Dr Barzah durrani, Sheikh Zayed Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Sheikh Zayed Medical College
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Choosing Better Drug Option for Sedation in Pediatric Population Intraoperatively
MeSH Terms: interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- midazola. (Experimental): Inj.midazolam
  Interventions: Drug: Midazolam
- Dexnedetomidine (Experimental): inj.dexmedetomidine
  Interventions: Drug: Dexmedetomidine injection

INTERVENTIONS:
Drug: Dexmedetomidine injection — Inj precedex 200mcg in 1ml given in stat doses
  Other Names: Precidex
  Arms: Dexnedetomidine
Drug: Midazolam — Inj.midazolam 5mg/5ml given in stat doses
  Arms: midazola.

SUMMARY:
Comparison of sedative effects of dexmedetomidine and midazolam using ramsay sedation scores intraoperatively in children undergoing inguinal hernia repair.

DETAILED DESCRIPTION:
a randomized controlled trial to compare the sesative effects of dexmedetomidine and midazolam in pediatric population planned for inguinal herna repair under TIVA in sheikh zayed hospital rahim yar khan.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II Age 6 to 12 years Any gender

Exclusion Criteria:

* ASA III and above Age less than 2 years and above 12 years Congenital heart disease Cardiac arrythmias Congenital abnormalities Respiratory disease Endocrine disorders Mental retardation Organ dysfunction Bleeding disorders Physician or family refusal Previous surgeries Allergy to any drug

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Dexmedetomidine is better sedative agent than midazolam in pediatric population | 25 minutes

SECONDARY OUTCOMES:
Midazolam is better sedating agent than dexmedetomidine in pediatric population | 25 minutes
Midazolam and dexmedetomidine are equally good sedating agents in pediatric population | 25 minutes

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From synopsis approval till completion of sample size